CLINICAL TRIAL: NCT00583466
Title: Evaluation of Blood as a Submucosal Cushion During Endoscopic Polypectomy and Mucosal Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00008376
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Large Polyps in the Gastrointestinal Tract
Keywords: submucosal cushion; polypectomy; endoscopic mucosal resection
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Normal saline arm (Active Comparator): Polypectomy with normal saline injected for submucosal cushion creation
  Interventions: Drug: Normal saline
- 2 HPMC arm (Active Comparator): Polypectomy after injection of hydroxypropyl methylcellulose (HPMC) to create submucosal cushion
  Interventions: Drug: HPMC
- 3 Blood arm (Experimental): Polypectomy after injection of autologous blood
  Interventions: Drug: Autologous blood injection

INTERVENTIONS:
Drug: Autologous blood injection — Autologous blood will be drawn from the patient and then reinjected under the lesion to create a safety cushion
  Arms: 3 Blood arm
Drug: Normal saline — Normal saline will be injected under the lesion to create submucosal cushion
  Arms: 1 Normal saline arm
Drug: HPMC — Hydroxypropyl methylcellulose (HPMC) will be injected under the lesion to create submucosal cushion
  Arms: 2 HPMC arm

SUMMARY:
For removal of large flat lesions of the gastro-intestinal tract injection of a solution under the lesion creates a "safety" cushion and protects from damage to the gastrointestinal tract wall. Various solutions are currently used, but some of them are easy to inject but quickly dissipate (normal saline),other solutions are more longer lasting (hydroxypropyl methylcellulose, hyaluronic acid, etc) but are very difficult to inject and can be expensive and not always available. The investigators performed previously animal experiments which demonstrated that blood is easy to inject and creates a protective cushion which lasts longer than other fluids which are currently used for protective cushion creation.

DETAILED DESCRIPTION:
For removal of large flat lesions of the gastro-intestinal tract injection of a solution under the lesion creates a "safety" cushion and protects from damage to the gastrointestinal tract wall. Various solutions are currently used, but some of them are easy to inject but quickly dissipate (normal saline),other solutions are more longer lasting (hydroxypropyl methylcellulose, hyaluronic acid, etc) but are very difficult to inject and can be expensive and not always available. The investigators decided to use blood drawn from the patient for injection under the lesion. The investigators performed previously animal experiments which demonstrated that blood is easy to inject and creates a protective cushion which lasts longer than other fluids which are currently used for protective cushion creation. Blood can also have local hemostatic action preventing from bleeding during polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* Polyps equal or larger than 1 cm

Exclusion Criteria:

* Coagulopathy
* Inability to sign informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V. Kantsevoy, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Giday SA, Magno P, Buscaglia JM, Canto MI, Ko CW, Shin EJ, Xia L, Wroblewski LM, Clarke JO, Kalloo AN, Jagannath SB, Kantsevoy SV. Is blood the ideal submucosal cushioning agent? A comparative study in a porcine model. Endoscopy. 2006 Dec;38(12):1230-4. doi: 10.1055/s-2006-944971. PMID 17163324

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No data on how participants were randomized, and no further baseline data (other than categorical age and sex) are available for this record. The PI has left the institution and has been contacted. Per the PI the data are no longer available and the study has not been published.
Groups:
- All Participants: Polypectomy with normal saline injected for submucosal cushion creation Normal saline: Normal saline will be injected under the lesion to create submucosal cushion
  OR
  Polypectomy after injection of hydroxypropyl methylcellulose (HPMC) to create submucosal cushion HPMC: Hydroxypropyl methylcellulose (HPMC) will be injected under the lesion to create submucosal cushion
  OR
  Polypectomy after injection of autologous blood Autologous blood injection: Autologous blood will be drawn from the patient and then reinjected under the lesion to create a safety cushion
Period: Overall Study
Arm/Group | All Participants
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No data on how participants were randomized, and no further baseline data (other than categorical age and sex) are available for this record. The PI has left the institution and has been contacted. Per the PI the data are no longer available and the study has not been published.
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Customized [Count of Participants; unit: Participants]
  >= 18, <= 90 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Duration of the Submucosal Cushion
Time Frame: Immediately after the procedure, Up to 5 minutes
Population: No data is available for this record. The PI has left the institution and has been contacted. Per the PI the data is no longer available and the study has not been published.
Arm/Group | 1 Normal Saline Arm | 2 HPMC Arm | 3 Blood Arm
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: There is no adverse event data available for this record. The PI has left the institution and has been contacted. Per the PI the data is no longer available and the study has not been published.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes